CLINICAL TRIAL: NCT03715413
Title: Analgesic Efficacy of Pulsed Radiofrequency in Non-cyclic Mastalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, lecturer of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansouraU3
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Breast Fibroadenoma
Keywords: pulsed radiofrequency, non-cyclic mastalgia
MeSH Terms: conditions — Fibroadenoma | interventions — Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen group (Other): they was received Tamoxifen 10 mg daily.
  Interventions: Drug: Tamoxifen
- Tamoxifen and pulsed radiofrequency group (Active Comparator): they was received Tamoxifen 10 mg daily and pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia.
  Interventions: Other: pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia.; Drug: Tamoxifen

INTERVENTIONS:
Other: pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia. — Patients were lying prone. Firstly, T2, 3, 4 disc level was detected then the target 2nd, 3rd and 4th thoracic nerve roots were identified. After marking the entry points, adequate sterilization of the skin was achieved using bovidone iodine then the skin was anasthesied by 2 ml lidocaine 2% at each entry point. The Baileys radio frequency (RF) 22G, 10 cm, sharp needles with 10 mm active tip was introduced to face the 2nd, 3rd and 4th thoracic nerve roots.The PRF course was carried out at 42°C for 120 s twice at each level followed by injection of 1 ml lidocaine 2% and 1 ml dexamethasone 4 mg at each level.
  Arms: Tamoxifen and pulsed radiofrequency group
Drug: Tamoxifen — received Tamoxifen 10 mg daily

SUMMARY:
Background: Breast pain, mastalgia or mastodynia, is recognized as an organic benign breast disease. Mastalgia may be bilateral, may be in only one breast or part of one breast, and may radiate to the axilla and down the medial aspect of the upper arm. This study aimed to evaluate the additional pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia to the routine regimen treatment of mastalgia tamoxifen 10 mg daily may improve breast pain severity and quality of life.

Method: Patients was randomly classified into two groups:Group A (n=13): they was received Tamoxifen 10 mg daily. Group B (n=13): they was received Tamoxifen 10 mg daily and pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia. The following parameters were monitored: Primary outcome: VAS after injection and at interval two weeks, 1, 2 and 3 months after injection. Secondary outcome:1-Immediate complications for ex. Hematoma, neurological deficits or respiratory insufficiency (dyspnea or pneumothorax).2-Need for analgesic intake was recorded.3-Side effect of Tamoxifen as nausea, vomiting, hot flashes and dizziness.4-Quality of life (The American Chronic Pain Association's Quality of life scale).

DETAILED DESCRIPTION:
Introduction:

Breast pain, mastalgia or mastodynia, is recognized as an organic benign breast disease . It can be severe enough to cause disturbances in normal quality of life rating which leads to disorders in sexual, physical, and social activities. When compared with other conditions, it will be similar to chronic cancer pain in the mean pain-index .

Breast pain is classified into three main categories: cyclical, non-cyclical and extra-mammary mastalgia. Cyclical pain is the commonest and it has a temporal association with the menstrual cycle. Pain characteristically starts in the days before menstruation and gradually increases. It tends to subside once menstruation has started and often disappears after a few days. Pain in these women usually abates after the menopause. These factors suggest a hormonal aetiology, high level of estrogen, low level of progesterone, and imbalance in estrogen to progesterone ratio are assumed among its causes, as well. Furthermore, many women associate the onset and resolution of cyclical mastalgia with a hormonal event, such as pregnancy or taking the oral contraceptive pill .

In contrast, there is no relationship to the menstrual cycle with non-cyclical mastalgia. Non-cyclic breast pain may result from pregnancy, mastitis, trauma, thrombophlebitis, macrocysts, psychologic disturbance, benign tumors, or cancer. However, only a minority of breast pain is explained by these conditions. Most non-cyclic breast pain arises for unknown reasons. Typically, it presents at a later age; most women are in the fourth or fifth decade of life at diagnosis. Many women are postmenopausal at onset of symptoms. Unfortunately, the course of both cyclical and non-cyclical mastalgia may be long and last many years.

The origin of extra-mammary pain is variable. Referred pain from cardiac, pulmonary and gastrointestinal causes, such as angina, pneumonia and oesophagitis, respectively, need to be excluded. A common cause of extra-mammary mastalgia arises from inflammation of the costochondral junctions of the chest wall (Tietze's disease). This condition usually resolves with rest and non-steroidal anti-inflammatory drugs .

Mastalgia may be bilateral, may be in only one breast or part of one breast, and may radiate to the axilla and down the medial aspect of the upper arm. The affected breast is often extremely tender to touch and pain may be accompanied by swelling and congestion.

A variety of medical therapies such as non-steroidal anti-inflammatory drugs (NSAIDs), vitamin B2, B6, E and C, diuretics, progesterone, thyroxin, Tamoxifen, Bromocriptine, Danazol, and plant extracts like evening primrose oil (EPO) and vitexagnus castus have been recommended for treatment of mastalgia. Unfortunately, Non-cyclic mastalgia responds poorly to medical treatment.

Psychological reassurance and active life style play a role to decrease the pain and low-fat, high-carbohydrate diet can also effect an improvement.

the female breast supplied its innervation from the anterior and lateral cutaneous branches of the second to the sixth intercostal nerves .

Tamoxifen is one of the medical treatment of mastalgia and considered as a first medication line. Tamoxifen 10 mg daily is effective in the treatment of mastalgia. It has side effects commonly observed in short-term treatment as weight gain, nausea, hot flashes (10%), bloating (5% or less), menstrual irregularity, amenorrhea (10%) and vaginal dryness. Thromboembolic is a rare but serious side effects of tamoxifen so it is contraindicated in women with a history of thromboembolic disease.

Pulsed radiofrequency (PRF) has recently been developed with widely usage by pain practitioners as alternative therapeutic technique for relief of chronic pain .

In our study, the investigators aim that the additional pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia to the routine regimen treatment of mastalgia tamoxifen 10 mg daily may improve breast pain severity and quality of life.

Our proposal: Is to find that pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia may improve breast pain severity and quality of life.

Aim of the work: This study aimed to evaluate the efficacy of additional pulsed radiofrequency (2nd , 3rd and 4th thoracic dorsal root ganglia) to the routine regimen treatment of mastalgia tamoxifen 10 mg daily.

Hypothesis: Management of non cyclic mastalgia is a challenging issue needing more appropriate method to reach the best result.

Recharge Gap: To our knowledge, there is a no researches discuss this issue and how to manage it in best way.

Patients and methods:

After approval of the local ethics committee (Mansoura university), twenty six patients complain from non-cyclic mastalgia aged from 18 to 60 with VAS > 4 was enrolled in this prospective study who were recruited from outpatient pain clinic in Oncology Center Mansoura University.

Sample size:

It was assessed using G-power analysis. Assuming α (type I error) = 0.05 and β (type II error) = 0.2 (power = 80 %) and effect size (δ) = 0.6 yielded a total sample size of 26.

Patients was randomly classified into two groups:

Group A (n=13): they was received Tamoxifen 10 mg daily. Group B (n=13): they was received Tamoxifen 10 mg daily and pulsed radiofrequency of 2nd , 3rd and 4th thoracic dorsal root ganglia.

Exclusion criteria: cyclical mastalgia, extra-mammary mastalgia patients refusal, suspicion of malignancy, acute inflammatory breast conditions, presence of polycystic ovarian diseases or cervical hyperplasia, pregnant patients and patients during lactation period, coagulopathy disorder, sepsis at the side of injection, history of thromboembolic disease, mental disorder and who was not willing or cannot finish the whole study, disturbed anatomy (congenital, traumatic, and postsurgical), which increase the intervention difficulty.

All patients in group B will inform about the procedure and its possible consequences. Written informed consent was obtained from all patients before the procedure.

Technique:

An intravenous cannula was inserted and secured. All suitable resuscitation equipment and drugs will available. Vital signs, heart rate, blood pressure and oxygen saturation will monitored throughout the procedure and up to 1 hour after the block performance.

Resuscitation equipment must be readily available including endotracheal tubes of different sizes, ambu bag, ventilator, druges eg. atropine and adrenaline.

The procedures were performed on a 64 MDCT scanner (Brilliance 64-Philips). The CT acquisition parameters were 200 mAs, 120 kVp, 512 × 512 matrix, 1.172 pitches, 64 × 0.625 mm section collimation, and 4 mm slice thickness.

Patients were lying prone. First, a level of T2, 3, 4 disc was detected then the target 2nd, 3rd and 4th thoracic nerve roots were identified. After marking the entry points, adequate sterilization of the skin was achieved using bovidone iodine then the skin was anasthesied by 2 ml lidocaine 2% at each entry point. The Baileys radio frequency (RF) 22G, 10 cm, sharp needles with 10 mm active tip was introduced to face the 2nd, 3rd and 4th thoracic nerve roots. If the lung or the pleura are within the needle path injection of saline in order to push the lung or the pleura away from the field.

When confirm the place of the needles tips, the sensory and motor stimulations were done by the RF generator to get sensory paresthesia along T2, T3 and T4 dermatomes at 0.4-0.8 V and intercostal fasciculation were obtained at double the sensory amplitude.

The PRF course was carried out at 42°C for 120 s twice at each level followed by injection of 1 ml lidocaine 2% and 1 ml dexamethasone 4 mg at each level.

After intervention, All patients were transferred to a recovery room for observation and record any complication.

ELIGIBILITY:
Inclusion Criteria:

* complain from non-cyclic mastalgia aged from 20 to 60 with VAS > 4

Exclusion Criteria:

* cyclical mastalgia
* extra-mammary mastalgia
* patients refusal
* suspicion of malignancy
* acute inflammatory breast conditions
* presence of polycystic ovarian diseases or cervical hyperplasia
* pregnant patients and patients during lactation period
* coagulopathy disorder
* sepsis at the side of injection
* history of thromboembolic disease
* mental disorder and who was not willing or cannot finish the whole study
* disturbed anatomy (congenital, traumatic, and postsurgical), which increase the intervention difficulty.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
VAS | 3 months
  0=no pain, 10=worst pain

SECONDARY OUTCOMES:
Immediate complications for ex | one day
  Hematoma, neurological deficits or respiratory insufficiency (dyspnea or pneumothorax).
Side effect of Tamoxifen | 3 months
  nausea, vomiting, hot flashes and dizziness.

CONTACTS AND LOCATIONS:
Locations (1):
- Yahay wahba, Al Mansurah, Egypt